CLINICAL TRIAL: NCT06172712
Title: COPD Exacerbation Modelling Study Using Daily-life Data From Unobtrusive Sensors - the TOLIFE Clinical Study A
Brief Title: COPD Exacerbation Modelling Using Unobtrusive Sensors - the TOLIFE Clinical Study A
Acronym: CSA
Status: Recruiting | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: University of Pisa (Other); LungenClinic Grosshansdorf (Other); Hospital del Mar Research Institute (Unknown); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Universidad Politecnica de Madrid (Other); TIMELEX (Unknown); Avvale (Unknown)
Responsible Party: Principal Investigator, Judith Garcia-Aymerich, Research Professor, Barcelona Institute for Global Health
Other Study IDs: 101057103CSA
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Exacerbation; Remote patient monitoring; Predictive modeling
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Variations in daily life activity signals detected by unobtrusive sensors — Patients will be equipped with unobtrusive devices for a duration of 12 months. Throughout this period, they will attend scheduled visits every three months following the baseline visit. These assessments will focus on determining the frequency of exacerbations, evaluating exercise capacity, measuring the severity of dyspnea, and assessing health-related quality of life. The data gathered from the sensors embedded in these unobtrusive devices will be instrumental in developing AI-based models. These models aim to accurately predict COPD exacerbations and effectively estimate the progression of the previously mentioned health outcome.

SUMMARY:
This work is a multicentric prospective cohort study designed to improve chronic obstructive pulmonary disease (COPD) treatment and management. The study involves 150 patients diagnosed with COPD who are at risk of exacerbations. These patients are recruited from three tertiary hospitals in Spain, Germany, and Italy. The study will last 18 months, with a 12-month follow-up duration for each patient. The primary objective of this study is to develop and test Artificial Intelligence (AI)-based models that can predict moderate-to-severe COPD exacerbations early on. This will be done by analyzing daily-life data collected from unobtrusive sensors that monitor patients' psycho-physiological and environmental signals. By accurately predicting exacerbations, the study aims to support clinicians in providing more precise, optimized, and personalized treatment to COPD patients. A secondary objective is to train and test AI-based models to estimate the 12-month dynamics of health-related quality of life (HRQoL) in COPD patients. This will involve analyzing data related to the patients' functional exercise capacity, dyspnea (difficulty breathing), and health-related quality of life, as measured by the Clinical COPD Questionnaire (CCQ) score and the COPD Assessment Test (CAT) score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (FEV1/FVC < 0.7) for at least a year.
* Participants with moderate-to-very severe COPD (FEV1 ≤ 80% predicted)
* Documented history of ≥ 1 moderate (treated with SABDs and oral corticosteroids ± antibiotics) or severe COPD exacerbation* within 12 months before enrolment.
* Adults aged 40 or over.
* Able to walk 4 meters independently with or without walking aids.
* Anticipated availability for repeated study visits over 12 months.
* Willingness to use smart sensors.
* Able to read and write in the first language in the respective location.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and the study protocol.

Exclusion Criteria:

* Occurrence of any of the following within three months before informed consent: myocardial infarction, hospitalization for unstable angina, stroke, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), implantation of a cardiac resynchronization therapy device (CRTD).
* Uncontrolled congestive heart disease (NYHA class >3).
* Having undergone major lung surgery (e.g., lung transplant)
* Primary respiratory diseases other than COPD.
* Participant who has experienced a major respiratory infection or exacerbation within 2 weeks before screening
* Lung volume reduction within six months before screening.
* Active treatment for cancer or other malignant diseases that in the opinion of the investigator, have an impact on the patient's quality of life such as to prevent adherence to the study.
* Acute psychosis or major psychiatric disorders or continued substance abuse.
* Severe disease that limits survival to 1 year.
* Patients with severe cognitive impairment (MMSE < 18).
* Substantial limitations in mobility due to factors other than COPD.
* Inability to follow the study procedures (e.g., due to language problems, psychological disorders) or unable to read, understand and fill in a questionnaire.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study targets COPD patients at risk of moderate-to-severe exacerbations. Participants will be recruited from three European tertiary care hospitals: Hospital del Mar in Barcelona, Spain; the Pulmonary Research Institute in Grosshansdorf, Germany; and Azienda Ospedaliera Universitaria Pisana in Pisa, Italy. Recruitment sources include research registers, hospital records, and referrals.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of moderate-to-severe COPD exacerbations | Months 3, 6, 9, and 12
  Occurrence of moderate-to-severe COPD exacerbations at months 3, 6, 9, and 12, through medical records

SECONDARY OUTCOMES:
Changes in the health-related quality of life | Baseline, Month 3, 6, 9 and 12
  Health-related quality of life at baseline, months 3, 6, 9, and 12, using the Clinical COPD Questionnaire (CCQ) and the COPD Assessment Test (CAT). The CCQ score ranges from 0 to 6, and the CAT score ranges from 0 to 40. Both questionnaires use higher scores to indicate a more severe impact of COPD on a patient's life.
Changes in the functional exercise capacity | Baseline, Month 3, 6, 9 and 12
  Changes in the functional exercise capacity at baseline, month 3, 6, 9 and 12, as measured by the Six-minute walking distance
Changes in the dyspnoea severity grade | Baseline, Month 3, 6, 9 and 12
  Changes in the dyspnoea severity grade at baseline, month 3, 6, 9, and 12, as measured by the modified Medical Research Council (MRC) Dyspnoea scale. The mMRC Dyspnoea scale ranges from 0 to 4, with higher scores indicating more severe dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Garcia-Aymerich, Principal Investigator — Barcelona Institute for Global Health
Locations (3):
- Pulmonary Research Institute, Großhansdorf, Schleswig-Holstein, Germany
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy
- Hospital del Mar Research Institute, Barcelona, Spain